CLINICAL TRIAL: NCT06204237
Title: Safety, Tolerability, and Biodistribution of [89Zr]Zr-DFO-APAC (Phase 0) in Subjects With Peripheral Arterial Occlusive Disease / Critical Limb Ischemia (PAOD/CLI) and Healthy Volunteers - an Open Label PET Study (Acronyms: 89Zr = Zirconium-89, DFO = Desferrioxamine, APAC = AntiPlatelet AntiCoagulant, PET/CT = Positron Emission Tomography/Computed Tomography)
Brief Title: Safety, Tolerability, and Biodistribution of [89Zr]Zr-DFO-APAC in Subjects With PAOD/CLI and Healthy Volunteers (Acronyms: 89Zr = Zirconium-89, DFO = Desferrioxamine, APAC = AntiPlatelet AntiCoagulant, PET/CT = Positron Emission Tomography/Computed Tomography)
Acronym: CHASE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aplagon Oy (Industry)
Collaborators: TRACER Europe BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-505287-11-01; 17489 (Registry Identifier: UMCG PaNaMa registry)
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Arterial Occlusive Disease; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [89Zr]Zr-DFO-APAC (Experimental)
  Interventions: Drug: [89Zr]Zr-DFO-APAC; Radiation: PET/CT scan

INTERVENTIONS:
Drug: [89Zr]Zr-DFO-APAC — All participants will receive a single i.v. injection of [89Zr]Zr-DFO-APAC 15 MBq (Megabecquerel).
Radiation: PET/CT scan — The IMP administration will be followed by whole-body PET/CT scanning (day 1), and repeated PET/CT scans on days 3 and 7.

SUMMARY:
The goal of this Phase 0 clinical trial is to evaluate safety and biodistribution of [89Zr]Zr-DFO-APAC in patients with peripheral arterial occlusive disease / critical limb ischemia (PAOD/CLI) and healthy volunteers. The main questions it aims to answer are:

* What is the safety, tolerability and pharmacokinetic profile (PK: both systemic and local vascular injury site-specific PK) of [89Zr]Zr-DFO-APAC?
* What is the biodistribution and internal radiation dosimetry of the tracer dose of [89Zr]Zr-DFO-APAC?
* What is the binding and retention time of [89Zr]Zr-DFO-APAC to arteries and atherosclerotic or microvascular lesions? Participants will receive a dose of the [89Zr]Zr-DFO-APAC (IMP) and PET/CT imaging is performed on days 1, 3 and 7, and follow-up visit 7-14 days post IMP dosing.

ELIGIBILITY:
INCLUSION CRITERIA PATIENTS

1. Males and females aged 40-85 years.
2. PAOD/CLI patients Rutherford categories 1-4 and category 5 with Wlfl wound grade of 0 or 1.
3. Estimated glomerular filtration rate (eGFR) >46 mL/min/1.73 m2 as per calculation of Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).
4. CT angiography with contrast agent performed of within 3 months of the patients' first PET-scan as part of diagnostics of PAOD, with results available in the subject's medical records.
5. No surgical or endovascular intervention for PAOD within 1 year of the first PET/CT-scan or planned between inclusion and the patients' last PET-scan.
6. Provision of valid informed consent and capability to communicate well with the investigator.
7. Pre-menopausal woman must be willing to practise highly effective contraception for 195 days after IMP administration.
8. Men must be willing to practise highly effective contraception for 105 days after IMP administration, including condom use during the first 15 days to prevent transmission of 89-Zr to a partner of childbearing potential.
9. Patients should be able to understand all study-related information in Dutch.

EXCLUSION CRITERIA PATIENTS

1. Acute limb-threatening ischemia (e.g., embolic disease).
2. An existing aneurysm that requires surgical intervention.
3. Medical history of, or condition known to be associated with impaired hemostasis, such as an increased intracranial bleeding risk e.g., previous history of intracranial hemorrhage, subarachnoidal bleeding, hemorrhagic stroke, or gastrointestinal or retroperitoneal bleeding, or any inherited or acquired bleeding disorder, such as von Willebrand disease or hemophilia.
4. Any cerebrovascular event (including transient ischemic attack, thrombotic or embolic stroke) within the past year.
5. Diagnosis of autoimmune (Type 1, or latent autoimmune diabetes in adults (LADA))diabetes mellitus.
6. HbA1c >10% at screening.
7. Current use of anticoagulant therapy (warfarin, apixaban, rivaroxaban, dabigatran, edoxaban, fondaparinux, or any heparin derivative) for any medical reason.
8. Patients treated with combined antiplatelet agents, excluding a single agent, such as acetylsalicylic acid (up to 100 mg QD) or clopidogrel (up to 75 mg QD).
9. Use of non-steroidal anti-inflammatory medications within 2 weeks prior to dosing with [89Zr]Zr-DFO-APAC. If pain relief is required, paracetamol may be used.
10. Use of selective serotonin reuptake inhibitor (SSRI) medications within 2 weeks prior to dosing with [89Zr]Zr-DFO-APAC.
11. Major surgery, major trauma or any endovascular intervention within the past 90 days or organ biopsy or diagnostic angiography within the past 30 days prior to the screening visit.
12. Uncontrolled arterial hypertension (persistent systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg).
13. Hemoglobin <8.0 mmol/L (130 g/l) (men) or <7.5 mmol/L (120 g/l) (women) at screening, or platelet count <150 x 109/L and leukocyte count >12 x 109/L.
14. Clinically significantly prolonged plasma prothrombin time (PT) and activated plasma partial thromboplastin time (APTT) (> 1.2-fold).
15. Patients with a medical history of heparin-induced thrombocytopenia.
16. Patients with known significant liver disease, incl. an alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) level > 2.5 x ULN (Upper limit normal) at screening.
17. A diagnosis of severe chronic kidney disease, defined as having a glomerular filtration rate (GFR) category 4 or 5 (GFR ≤ 45 mL/min/1.73 m2) and albuminuria stage A3 albumin:creatinine ratio (ACR) of >300 mg/g).
18. Patients with an active malignancy or who have received treatment for any malignancy within 1 year before the screening visit, except for localized basal cell or squamous cell skin cancer that has been cured at least 90 days before screening.
19. Patients with a history of metastatic malignancy.
20. Women who are pregnant or lactating.
21. Patients with a known allergy or hypersensitivity to heparin or heparin products, and/or antiplatelet agents (e.g., aspirin or clopidogrel).
22. Participation in an investigational drug or device study within 30 days prior to screening.
23. Patients who have ever received treatment with an antibody or gene therapy product or participated in a clinical trial with such agents (unless there is evidence that they received placebo only).
24. Patients with known antiphospholipid antibody syndrome or other thrombophilia.
25. Patients with a medical history of severe infection or vasculitis due to an autoimmune disease, inflammatory bowel disease (IBD) or Crohn's disease.
26. Any concomitant disease or condition that could interfere with, or the treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject.
27. Patients unable or unwilling to comply with the protocol or to cooperate fully with the investigator or site personnel.
28. Patients with anamnestic history of drug abuse (defined as illicit drug use) or anamnestic history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within the past 12 months.

INCLUSION CRITERIA HEALTHY VOLUNTEERS

1. Male or female volunteers 40-80 years old, inclusive.
2. Healthy status defined by the absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, serology and urinalysis.
3. No diagnosis of diabetes, pre-diabetes or insulin resistance.
4. Normal eGFR as per calculation of Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).
5. Premenopausal woman must be willing to practise highly effective contraception for 195 days after IMP administration.
6. Men must be willing to practise highly effective contraception for 105 days after IMP administration, including condom use during the first 15 days to prevent transmission of 89-Zr to a partner of childbearing potential
7. Healthy volunteers should be able to understand all study-related information in Dutch.

EXCLUSION CRITERIA HEALTY VOLUNTEERS

1. Any sign or symptom of PAOD/CLI or other cardiovascular disease.
2. Abnormal ankle-brachial index (ABI) at rest and/or decrease of ABI following treadmill exercise.
3. Use of any anticoagulant or antiplatelet (not including aspirin at recommended doses) agent within the recent 12 months before screening.
4. Any regular prescription or over-the-counter medication, except for vitamins.
5. Medical history of heparin-induced thrombocytopenia.
6. Medical history of atrial fibrillation and/or those with a mechanical heart valve.
7. Major surgery, major trauma or organ biopsy within the past 90 days before screening.
8. Medical history of, or any condition, associated with an increased bleeding risk.
9. Arterial hypertension (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg.
10. Subjects with a medical history of, or an existing aneurysm.
11. Hemoglobin <8.0 mmol/L (130 g/l) (men) or <7.5 mmol/L (120 g/l) (women) at screening or platelet count < 150 x 109/L or leukocyte count above normal (12 x 109/L).
12. Clinically significantly prolonged prothrombin time (PT) and activated partial thromboplastin time (APTT) (> 1.2-fold).
13. Participation in an investigational drug or device study within 30 days prior to screening.
14. Subjects who have ever received treatment with an antibody or gene therapy product or participated in a clinical trial with such agents (unless there is evidence that they were received placebo only).
15. Subjects with known thrombophilia.
16. Women who are pregnant or lactating.
17. Subjects unable or unwilling to comply with the protocol or to cooperate fully with the investigator or site personnel.
18. Subjects with anamnestic history of drug abuse (defined as illicit drug use) or a anamnestic history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within the past 3 months.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (AE) (safety and tolerability) | Study duration (Up to 21 days)
  Occurrence and severity of one or more treatment-emergent AEs from the time of i.v. administration of [89Zr]Zr-DFO-APAC until the end of the follow-up period, and changes in plasma/serum clinical chemistry, hematology, coagulation variables, vital signs, ECG, and physical examination findings.

OTHER OUTCOMES:
Biodistribution and radiation dosimetry of [89Zr]Zr following administration of [89Zr]Zr-DFO-APAC | Day 1, day 3 and day 7 after dosing
  Dosimetry estimates and cumulated radioactivity exposure by source region and the entire body in the first three participants including analysis of radioactivity in venous blood.

CONTACTS AND LOCATIONS:
Overall Officials: Schelto Kruijff, MD, Prof, Principal Investigator — University Medical Center Groningen, NL
Locations (1):
- The University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No